CLINICAL TRIAL: NCT04127916
Title: Bendamustine Plus Rituximab for Mantle Cell Lymphoma: a Multicenter Retrospective Analysis(BR-MCL)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Won Seog Kim, MD,phD,Division of hematology, Department of medicine, Samsung Medical Center
Other Study IDs: 2019-07-091
Record Dates: First submitted 2019-10-13; First posted 2019-10-16 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — Bendamustine Hydrochloride; Rituximab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Bendamustine — To investigate the efficacy and safety of bendamustine plus rituximab in patients with mantle cell lymphoma.
  Other Names: Rituximab

SUMMARY:
This study with retrospective data collection does not entail sample size calculation. The study will involve patients who received bendamustine + rituximab for relapsed/refractory mantle cell lymphoma and meet the inclusion/exclusion criteria at each participating study site. Considering the incidence of mantle cell lymphoma in Korea and the number of participating sites, the expected sample size is approximately 40.

DETAILED DESCRIPTION:
1. Inclusion criteria : Patients newly diagnosed with mantle cell lymphoma by a pathologist (based on the 2016 revision of the WHO classification) 1) mantle cell lymphoma 2) leukemic non-nodal mantle cell lymphoma 3) in situ mantle cell neoplasia
2. Age ≥ 19 years
3. Patients who received bendamustine + rituximab as initial therapy and patients who received bendamustine + rituximab for the treatment of relapsed/refractory condition are both included.

2. Exclusion criteria :

1. Patients whose clinical and pathological data are not available
2. Patients who were not treated with a combination of bendamustine and rituximab

Data of patients who received bendamustine + rituximab for relapsed/refractory mantle cell lymphoma collected before the date of first submission of an IRB application for new project will be analyzed.

The aim is to publish the data analysis and study results before December 2020. The expected overall study period is until December 2020.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients newly diagnosed with mantle cell lymphoma by a pathologist (based on the 2016 revision of the WHO classification)

  1. mantle cell lymphoma
  2. leukemic non-nodal mantle cell lymphoma
  3. in situ mantle cell neoplasia 2. Age ≥ 19 years 3. Patients who received bendamustine + rituximab as initial therapy and patients who received bendamustine + rituximab for the treatment of relapsed/refractory condition are both included.

Exclusion Criteria:

* 1. Patients whose clinical and pathological data are not available 2. Patients who were not treated with a combination of bendamustine and rituximab

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study with retrospective data collection does not entail sample size calculation. The study will involve patients who received bendamustine + rituximab for relapsed/refractory mantle cell lymphoma and meet the inclusion/exclusion criteria at each participating study site. Considering the incidence of mantle cell lymphoma in Korea and the number of participating sites, the expected sample size is approximately 40.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-01-30 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate, | 2020.12.30
  Overall response rate, including complete response and partial response

SECONDARY OUTCOMES:
Progression-free survival | 2020.12.30
  The length of time during and after the treatment of a disease, such as cancer, that a patient lives with the disease but it does not get worse
Overall survival | 2020.12.30
  The percentage of people in a study or treatment group still alive for a given period of time after diagnosis
Duration of response | 2020.12.30
  Duration of response
Treatment-emergent adverse event | 2020.12.30
  Treatment-emergent adverse event
Prognostic factor | 2020.12.30
  Prognostic factor

CONTACTS AND LOCATIONS:
Overall Officials: Kim wonseog, Professor, Principal Investigator — Samsung Medical Center
Locations (2):
- South Korea (2):
  - Samsung Medical Center, 81 Irwon-ro, Gangnam-gu, Seoul, Republic of Korea, Seoul
  - Samsung Medical Center, 81, Irwon-ro, Gangnam-gu, Seoul, Republic of Korea, Seoul

IPD SHARING:
Plan to Share IPD: No
There is no IPD sharing plan